CLINICAL TRIAL: NCT00633347
Title: Use of Antagonist Versus Agonist GnRH in Oocyte Recipient Endometrium Preparation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Carmina Vidal, MD, Gynaecologist IVI valencia; Principal Investigator, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VLC-CV-1006-02
Record Dates: First submitted 2008-02-21; First posted 2008-03-12 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Infertility
Keywords: oocyte donation; endometrial preparation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): A: Antagonist
  Interventions: Drug: Antagonist GnRH Cetrotide; Drug: Agonist GnRH Acetate Triptoreline
- B (Active Comparator): Agonist GnRH
  Interventions: Drug: Agonist GnRH Acetate Triptoreline

INTERVENTIONS:
Drug: Antagonist GnRH Cetrotide — Cetrotide 0.25 mg. daily/ 7 days
  Arms: A
Drug: Agonist GnRH Acetate Triptoreline — Acetate Triptorelina (Agonist GnRH), 3.75 mg. single dose

SUMMARY:
Oocyte donation is a well established procedure in assisted reproduction treatments (ART). It is demonstrated that the use of hormonal substitution therapy, for the synchronization of the cycles between the recipients and the donors, provides good results, similar to the ones obtained with the natural cycle. In the patients - recipients with preserved ovarian function, the recipient's natural cycle is annulled, thus preventing the spontaneous Luteinizing Hormone surge. Simultaneously and while waiting for the suitable donor, her endometrium is prepared. When the donation occurs and fertilization with the husband sperm takes place, her cycle is stimulated again in order to synchronize her window of implantation with the donor's ovulation.

Two different medications are commonly used to inhibit spontaneous ovulation: either GnRHa agonist or GnRH antagonists. The present study consists of the comparison between the single dose GnRH agonist (Decapeptyl 3,75 IM) and the 7 day dosage of GnRH antagonist (Cetrotide 0,25 mg). The administration of GnRHa is used fundamentally as a long liberation formulation, administered in a single intramuscular injection (IM), which is more practical in terms of use. Nevertheless, the unnecessary persistence and the potentially unfavorable action of GnRHa during the luteal phase and early gestation have questioned its use. The recovery of the Hypophysarian function begins only 8 weeks after the single injection of long liberation of triptorelina 3.75 mg. The GnRH antagonist (Cetrotide 0,25 mg) makes the hypofisary inhibition shorter than with the analogues and can prepare similar endometrium characteristics as a natural cycle. The recipients will be assigned randomly to a group of treatment or another.

ELIGIBILITY:
Inclusion Criteria:

* infertile females with preserved gonadal function
* ages 18 - 43 years old

Exclusion Criteria:

* BMI: > 28
* recurrent miscarriages
* severe male factor
* important miomas
* > 44 years old

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 570 (Actual)
Dates: Start 2007-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 1 month

SECONDARY OUTCOMES:
implantation rate | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Valencia, Valencia, Spain